CLINICAL TRIAL: NCT05521256
Title: A First Human Dose Study Investigating Safety, Tolerability, and Pharmacokinetics of Oral Single Doses of NNC0113-6856 in Healthy Male Participants
Brief Title: A Research Study of a New Medicine NNC0113-6856 in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9904-4825; U1111-1270-0813 (Other: World Health Organization (WHO)); 2021-005397-26 (EudraCT Number)
Record Dates: First submitted 2022-08-27; First posted 2022-08-30 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- NNC0113-6856 (Oral Cohort) (Experimental): Participants will receive single oral dose of NNC0113-6856 tablets in dose escalated manner.
  Interventions: Drug: NNC0113-6856
- Placebo (Placebo Comparator): Participants will receive single oral dose of placebo (NNC0113-6856) tablets in dose escalated manner.
  Interventions: Drug: Placebo
- NNC0113-6856 (i.v. Cohort) (Experimental): Participants will receive single dose of 1.5 milligrams (mg) NNC0113-6856 intravenously (i.v.).
  Interventions: Drug: NNC0113-6856

INTERVENTIONS:
Drug: NNC0113-6856 — Participants will receive NN0113-6856 orally or intravenously.
  Arms: NNC0113-6856 (Oral Cohort); NNC0113-6856 (i.v. Cohort)
Drug: Placebo — Participants will receive matching placebo of NNC0113-6856 for each of the oral cohorts.
  Arms: Placebo

SUMMARY:
In this study NN0113-6856 will be given to humans for the first time. We will be looking into how safe different single doses of the new investigational product NNC0113-6856 is and we will measure its amount as well as the amount of specific parts of the new investigational product in blood. The study will look at the effects of different single doses of NNC0113-6856. This could either be as an oral dose (cohort 1 to 5) or one injection into the vein (intravenous [IV]-cohort). Participant will get the investigational product either as one or two tablets (oral dose in cohort 1 to 5) or as injection into the vein (IV cohort). The study will last for about 6-10 weeks (up to 14 weeks in case of rescheduling for stand-by participants).

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index between 20.0 and 27.0 kilogram per meter square (kg/m^2)(both inclusive).

Exclusion Criteria:

* Glycated haemoglobin (HbA1c) greater than or equal to (>=) 6.5 percent (%) (48 millimoles per moles [mmol/mol]) at screening.
* Use of tobacco and nicotine products, defined as any of the below:

  * Smoking more than 5 cigarettes or the equivalent per day.
  * Not willing to refrain from smoking and use of nicotine substitute products during the inpatient periods.
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs or nutrients, as judged by the investigator.
* History of major surgical procedures involving the stomach potentially affecting absorption of trial products (example: subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery) or current presence of gastrointestinal implant
* Presence or history of pancreatitis (acute or chronic).
* Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.
* Any of the below laboratory safety parameters at screening outside the below laboratory range, see "Log of laboratory ranges used for laboratory parameter exclusion criterion" for specific values:

  * Alanine Aminotransferase (ALT) greater than (>) upper normal limit (UNL)
  * Aspartate aminotransferase (AST) > UNL
  * Bilirubin > UNL
  * Creatinine > UNL
  * International normalized ratio (INR) > UNL
* Precence or history of hepatitis

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | From time of dosing (day 1) until completion of the follow-up visit (Day 42)
  Measured as number of events.

SECONDARY OUTCOMES:
For oral cohorts- AUC0-tz,sema,single dose (SD): Area under the semaglutide plasma concentration-time curve from time 0 to tz after a single dose, where tz is the time of last quantifiable concentration | From pre-dose (day 1) to completion of follow-up visit (Day 42)
  Measured in hours*nanomoles per liter (h*nmol/L).
For oral cohorts- AUC0-infinity (∞),sema,SD: Area under the semaglutide plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) to completion of follow-up visit (Day 42)
  Measured in hours*nanomoles per liter (h*nmol/L).
For oral cohorts- Cmax,sema,SD: Maximum observed plasma concentration of semaglutide after a single dose | From pre-dose (day 1) to completion of follow-up visit (day 42)
  Measured in nanomoles per liter (nmol/L).
For oral cohorts- tmax,sema,SD: Time to maximum observed concentration of semaglutide after a single dose | From pre-dose (day 1) to completion of follow-up visit (day 42)
  Measured in hours (h).
For oral cohorts- t½,sema,SD: Terminal half-life of semaglutide after a single dose | From pre-dose (day 1) to completion of follow-up visit (day 42)
  Measured in hours (h).
For oral cohorts- AUC0-tz,6856,SD: Area under the NNC0113-6856 plasma concentration-time curve from time 0 to tz after a single dose, where tz is the time of last quantifiable concentration | From pre-dose (day 1) to completion of visit 5 (day 22)
  Measured in hours*nanomoles per liter (h*nmol/L).
For oral cohorts- AUC0-∞,6856,SD: Area under the NNC0113-6856 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) to completion of visit 5 (day 22)
  Measured as hours*nanomoles per liter (h*nmol/L).
For oral cohorts- Cmax,6856,SD: Maximum observed plasma concentration of NNC0113-6856 after a single dose | From pre-dose (day 1) to completion of visit 5 (day 22)
  Measured as nanomoles per liter (nmol/L).
For oral cohorts- tmax,6856,SD: Time to maximum observed concentration of NNC0113-6856 after a single dose | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in hours (h).
For oral cohorts- t½,6856,SD: Terminal half-life of NNC0113-6856 after a single dose | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in hours (h).
For oral cohorts- AUC0-tz,4768,SD: Area under the NNC0113-4768 plasma concentration-time curve from time 0 to tz after a single dose, where tz is the time of last quantifiable concentration | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in hours*nanomoles per liter (h*nmol/L).
For oral cohorts- AUC0-∞,4768,SD: Area under the NNC0113-4768 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in hours*nanomoles per liter (h*nmol/L).
For oral cohorts- Cmax,4768,SD: Maximum observed plasma concentration of NNC0113-4768 after a single dose | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in nanomoles per liter (nmol/L).
For oral cohorts- tmax,4768,SD: Time to maximum observed concentration of NNC0113-4768 after a single dose | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in hours (h).
For oral cohorts- t½,4768,SD: Terminal half-life of NNC0113-4768 after a single dose | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in hours (h).
For intravenous (i.v.) cohort- AUC0-infinity (∞),sema,SD: Area under the semaglutide plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) to completion of follow-up visit (day 42)
  Measured in hours*nanomoles per liter (h*nmol/L).
For i.v. cohort- t½,sema,SD: Terminal half-life of semaglutide after a single dose | From pre-dose (day 1) to completion of follow-up visit (day 42)
  Measured in hours (h).
For i.v. cohort- Cmax,sema,SD: Maximum observed plasma concentration of semaglutide after a single dose | From pre-dose (day 1) to completion of follow-up visit (day 42)
  Measured in nanomoles per liter (nmol/L).
For i.v. cohort- AUC0-∞,6856,SD: Area under the NNC0113-6856 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) to completion of visit 5 (day 22)
  Measured as hours*nanomoles per liter (h*nmol/L)
For i.v. cohort- t½,6856,SD: Terminal half-life of NNC0113-6856 after a single dose | From pre-dose (day 1) to completion of visit 5 (day 22)
  Measured in hours (h).
For i.v. cohort- CL6856,SD: Total plasma clearance of NNC0113-6856 after a single dose | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in liters per hour (L/h).
For i.v. cohort- Vz6856,SD: Apparent volume of distribution of NNC0113-6856 after a single dose based on plasma concentration values | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in liters (L).
For i.v. cohort- MRT6856,SD: Mean residence time for NNC0113-6856 after a single dose | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in hours (h).
For i.v. cohort- AUC0-infinity (∞),4768,SD: Area under the NNC0113-4768 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in hours*nanomoles per liter (h*nmol/L).
For i.v. cohort- t½,4768,SD: Terminal half-life of NNC0113-4768 after a single dose | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in hours (h).
For i.v. cohort and oral cohort- AUC0-∞,6856,SD/dose: Area under the NNC0113-6856 plasma concentration-time curve from 0 to infinity after a single dose divided by the dose administered | From pre-dose (day 1) to completion of visit 5 (Day 22)
  Measured in hours*nanomoles per liter per milligram (h*nmol/L/mg).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (3):
- Germany (3):
  - Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia
  - Profil GmbH & Co. KG, Mainz
  - Profil Institut für Stoffwechselforschung GmbH, Neuss

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com